CLINICAL TRIAL: NCT01053637
Title: Randomized Control Trial of Oral Narcotic Medication for Pain and Anxiety Management During Laceration Repair in the Pediatric Emergency Department
Brief Title: Pain and Anxiety Management With Oral Narcotic for Pediatric Suture Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Corrie Chumpitazi, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-22684
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Children; Lacerations; Procedures; Child; Pain
Keywords: lacerations; sutures; pediatrics; child; pain; Anxiety
MeSH Terms: conditions — Lacerations; Pain; Anxiety Disorders | interventions — oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocodone/acetaminophen (Experimental): Patients will receive 0.17 mg/kg hydrocodone component to a max of 10 mg hydrocodone.
  Interventions: Drug: hydrocodone/acetaminophen
- Sugar water (Placebo Comparator): Placebo
  Interventions: Drug: Sugar water

INTERVENTIONS:
Drug: hydrocodone/acetaminophen — 0.17 mg/kg hydrocodone component to max of 10 mg. If dose is vomited within 5 minutes, second dose may be administered.
  Other Names: Lortab; Vicodin
  Arms: Hydrocodone/acetaminophen
Drug: Sugar water — An equal volume of sugar water will be dispensed, as for the weight based 0.17 mg/kg hydrocodone solution given for the study drug
  Arms: Sugar water

SUMMARY:
The purpose of this study is:

* To determine whether oral narcotic medication versus placebo improves the pain and anxiety scores for pediatric patients requiring laceration repair in the pediatric emergency department and receiving the standard of care with lidocaine treatment
* To evaluate for a statistical difference in pain scores in children during laceration repair
* To evaluate for a statistical difference in State-Trait Anxiety Inventory for Children (STAIC) scores during laceration repair

DETAILED DESCRIPTION:
A prospective, double-blind, placebo-controlled, randomized clinical trial in a tertiary care pediatric emergency department with an annual census of 80,000 visits per year. Patients will be randomized by a randomization table with block randomization in the pharmacy to the oral narcotic or placebo group, and the pharmacist will be the only person aware of the randomization status of the patient. Allocation concealment will be ensured by opaque, sealed envelopes kept in the Emergency Department Pharmacy. Guardians of patients age 2 to 17 years of age will be consented for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 17 years
* Laceration of the skin and/or subcutaneous tissue requiring sutures
* American Society of Anesthesiologists (ASA) score of I or II

Exclusion Criteria:

* Major injuries in addition to laceration (suspected fracture, intracranial, intrathoracic, or intraabdominal bleeding or organ injury)
* Abnormal neurologic examination (such as head injury)
* Severe congenital heart disease
* Pregnancy
* Known opiate or acetaminophen allergy
* Require conscious sedation
* Have had narcotic or acetaminophen administration within 4 previous hours

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrie Chumpitazi, MD, Principal Investigator — Texas Childrens Hospital
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocodone/Acetaminophen | Sugar Water
Started | 43 | 42
Completed | 43 (2 with incomplete pain scores) | 42 (4 incomplete pain scores 4 proceeded to procedural sedation)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Hydrocodone/acetaminophen suspension (taste/color-matched)
- Placebo: Sugar solution
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5.25 [3.75 to 6.74] | 4.87 [3.57 to 6.27] | 5.1 [3.6 to 6.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 23
  Male | 36 | 26 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 12 | 8 | 20
  Caucasian | 4 | 10 | 14
  Hispanic | 25 | 23 | 48
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: Statistical Difference in Pain Scores in Children During Laceration Repair Between Study and Placebo Group
Description: Children's Hospital of Eastern Ontario Pain Scale, for children 2-7 years. This score ranks 6 categories: Cry, Facial expression, Verbal Response, Torso movement, Touch, and Leg movement. The scale varies by each category from 0-2 or 1-2 or 1-3; such that a minimum score is 4 (no pain) and a maximum score is 13 signifying greatest pain. This results in a 10 point scale of possible results, and is rated by an objective observer; the child life specialist at the bedside during the laceration repair. If the procedure was completed, there were no scores recorded at that time point.
Time Frame: 5 minutes
Population: The 2-7 year old population at primary outcome time point of 5 minutes. This 2-7 year old population: randomized 25 in each arm (50 total) but 5 had missing pain scores due to child life specialist availability at the time of repair. Older population had 35 patients enrolled, but 1 in the placebo group was excluded for missing pain scores.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Hydrocodone/Acetaminophen | Sugar Water
Number analyzed (Participants) | 23 | 22
units on a scale | 5 [4 to 6.5] | 7 [5.25 to 10]
Statistical Analysis 1: Comparison: Hydrocodone/Acetaminophen vs Sugar Water; Children's Hospital of Eastern Ontario Pain Scale, for children 2-7 years. This score ranks 6 categories: Cry, Facial expression, Verbal Response, Torso movement, Touch, and Leg movement. The scale varies by each category from 0-2 or 1-2 or 1-3; such that a minimum score is 4 (no pain) and a maximum score is 13 signifying greatest or worst pain; Test type: Superiority; p = 0.05, Fisher Exact — Pain at 5 minutes using Children's Hospital of Eastern Ontario Pain Scale validated in the younger population. Using a 2-point difference in CHEOPS pain scale as a clinically significant change, 34 patients were required in the younger 2- to 7 group

2. Secondary Outcome: Statistical Difference in State-Trait Anxiety Inventory for Children (STAIC) Scores for Children Aged 8-17 Years During Laceration Repair and VAS Pain Scale
Description: State-Trait Anxiety Inventory for Children - 20 questions with 3 answer options for each question.
  Scores range from 20 to 60 for state and 20 to 60 for trait with 60 being the higher (more or worse) anxiety on self-assessment. The VAS pain Scale from 0-10 was included in this older population as well.
Time Frame: 1 hour approximately (survey was given pre and post procedure so from 15 minutes to 1 hour after initial survey (or 5 minutes to 45 minutes after the procedure).
Population: State-Trait Anxiety Inventory for Children (STAIC) which is a 20 question tool, low score no anxiety and high score more anxiety. This test was only used for the 34 patients in the >7 years (8-17 years) category as this scale is validated in that population. The VAS Pain score was measured as well.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Hydrocodone/Acetaminophen | Sugar Water
Number analyzed (Participants) | 18 | 16
units on a scale
  State Anxiety Pre-Test | 34.5 [31.0 to 40.75] | 38.0 [32.5 to 41.75]
  State Anxiety Post-Test | 26.0 [24.0 to 30.0] | 29.0 [21.50 to 32.50]
  VAS Pain Score at 5 minutes | 0.1 [0.0 to 4.23] | 0.5 [0.0 to 1.2]
Statistical Analysis 1: Comparison: Hydrocodone/Acetaminophen vs Sugar Water; State-Trait Anxiety Inventory for Children pre vs. post procedure for matched pairs. Higher numbers indicated higher state anxiety. State Trait Anxiety Inventory for Children (STAIC) scores pre vs. post procedure for matched pairs. A lower STAIC score indicates less anxiety and a greater score indicates more anxiety based on Likert-type scales and analyzed using nonparametric testing; Test type: Other; p = 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Visual Analog Scale (VAS) Pain Score for Children > 7 Years.
Description: Visual Analog Scale from 0-10 as marked on a 10 cm line. 0 no pain, 10 worst pain.
  A child >7 group marks their pain on the line, and a mm measurement is made. Power based on a change in the Visual Analog Scale (VAS) for children > 7 years. A change in pain score of 10 mm (95% Confidence Interval 7-12 mm) was considered to be clinically significant based upon a previous study.
Time Frame: 30 minutes
Population: 1 placebo (sugar water) patient required sedation and 1 placebo (sugar water) patient had missing pain scores, so 14 patients for analysis. For the hydrocodone/acetaminophen group, baseline VAS score was not available for 1 participant. If the procedure was completed, there were no scores recorded at that time point (i.e. 20 minutes).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydrocodone/Acetaminophen | Sugar Water
Number analyzed (Participants) | 17 | 14
score on a scale
  Baseline | 0.5 [0.0 to 5.30] | 0.85 [0.0 to 4.85]
  5 minutes: number analyzed (Participants) | 17 | 13
  5 minutes | 0.1 [0.0 to 4.23] | 0.5 [0.0 to 1.20]
  10 minutes: number analyzed (Participants) | 17 | 10
  10 minutes | 0.0 [0.0 to 2.00] | 0.0 [0.0 to 1.60]
  15 minutes: number analyzed (Participants) | 12 | 4
  15 minutes | 0.0 [0.0 to 3.18] | 0.0 [0.0 to 0.75]
  20 minutes: number analyzed (Participants) | 0 | 0
  Procedure Finish: number analyzed (Participants) | 15 | 11
  Procedure Finish | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment through hospital discharge for the specific emergency department visit during which the patient was enrolled, and chart reviewed for return visit up to 72 hours from discharge.
Description: Any adverse event was reported directly to the study PI.
Arm/Group | Hydrocodone/Acetaminophen | Sugar Water
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes